CLINICAL TRIAL: NCT06008483
Title: A Dose Finding Study of CycloSam® (153-Sm-DOTMP) to Treat Solid Tumor(s) in the Bone or Metastatic to the Bone (Metastatic Prostate, Breast, and Lung, Osteosarcoma, Ewing's Sarcoma, and Other Solid Tumor(s) to the Bone All Eligible)
Brief Title: A Dose Finding Study to Treat Bone Tumor(s)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: QSAM Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: QSAM-001
Record Dates: First submitted 2023-08-04; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Bone Cancer; Bone Tumor; Solid Tumor; Metastatic Cancer to the Bone; Metastatic Tumor to the Bone
Keywords: Bone cancer; Bone Tumor; Solid Tumor; Metastatic Cancer to the Bone; Metastatic Tumor to the Bone
MeSH Terms: conditions — Bone Neoplasms

STUDY DESIGN:
Masking Description: This clinical trial is unblinded, non-randomized, and there is no placebo group. All participants receive active drug product.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Level 1 (Other): Everyone gets a first dose of 0.5 mCi/kg dose and then in 7 days a second dose of 0.5 mCi/kg
  Interventions: Drug: 153-Sm-DOTMP (Samarium-153-DOTMP)
- Dose Level 2 (Other): Everyone gets a first dose of 0.5 mCi/kg dose and then in 7 days a second dose of 1.0 mCi/kg
  Interventions: Drug: 153-Sm-DOTMP (Samarium-153-DOTMP)
- Dose Level 3 (Other): Everyone gets a first dose of 0.5 mCi/kg dose and then in 7 days a second dose of 2.0 mCi/kg
  Interventions: Drug: 153-Sm-DOTMP (Samarium-153-DOTMP)
- Dose Level 4 (Other): Everyone gets a first dose of 0.5 mCi/kg dose and then in 7 days a second dose of 3.0 mCi/kg
  Interventions: Drug: 153-Sm-DOTMP (Samarium-153-DOTMP)

INTERVENTIONS:
Drug: 153-Sm-DOTMP (Samarium-153-DOTMP) — This is an open-label, unblinded, multi-center, dose-finding study of 153Sm-DOTMP (CycloSam®) to identify the MTD of 153Sm- DOTMP, given as a tandemly administered pair of doses to subjects with solid tumors visible on bone scan.

SUMMARY:
To determine the Maximum Tolerated Dose (MTD) of CycloSam®, Samarium-153-DOTMP (Sm-153-DOTMP), a radiopharmaceutical that delivers radiation to the bone when injected, given as a tandemly administered pair of doses to subjects with one or more solid tumor(s) in the bone or metastatic solid tumors to the bone that are visible on bone scan.

DETAILED DESCRIPTION:
This is an open-label, unblinded, multi-center, dose-finding study of 153-Sm-DOTMP (CycloSam®), a radiopharmaceutical that delivers radiation to the bone when injected, to identify the MTD of 153-Sm- DOTMP, given as a tandemly administered pair of doses to subjects with solid tumors visible on bone scan. The MTD will be defined as the dose level that produces a dose limiting toxicity (DLT) rate no greater than 25%. DLTs will be defined as any grade 3 or greater hematologic or nonhematologic toxicity, as defined by the National Cancer Institute (NCI) - Common Terminology Criteria for Adverse Events (CTCAE), experienced during a 42 day observation window. Clinical response will be defined as either stable disease (SD) or a decrease in the size of the tumor by radiographic imaging (which may include computed tomography [CT] or magnetic resonance imaging [MRI]) using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.The Day 1 dose will remain constant at 0.5 mCi/kg, with the Day 8 dose escalated from 0.5 mCi/kg (dose level 1) to 1.0 mCi/kg (dose level 2) to 2.0 mCi/kg (dose level 3) and then to 3.0 mCi/kg (dose level 4).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will be between the ages of 15 and 75, inclusive.
2. Subjects must have a histologically confirmed diagnosis of a solid tumor metastatic to bone, or a histologically confirmed diagnosis of a solid tumor to the bone or metastatic to the bone.
3. Subjects must have measurable disease on anatomic imaging that is also avid for phosphonate compounds as demonstrated by a positive 99mTc diphosphonate bone scan. Not all lesions must be positive on bone scan.
4. Adequate organ function, including:

   i. Adequate renal function, defined as a measured creatinine clearance >70 mL/min/1.73 m2 or normal radioisotope glomerular filtration rate (GFR).

   ii. Adequate hematologic function, defined as a platelet count >100,000 cells/mm3 and an absolute neutrophil count (ANC) >1,000 cells/mm3.
5. Life expectancy of at least eight weeks.
6. Karnofsky performance status >50%.
7. Subjects must have adequately recovered from the effects of any prior chemotherapy, as determined by the treating physician and study team, based in part on organ function defined above. Toxicities from previous therapies must have recovered to CTCAE v5.0 grade ≤1. Subjects with Grade 2 anemia per CTCAE v5.0 will be permitted as long as the subject has normal cardiac function.
8. Adequate cardiac function. Subjects with previously identified cardiac disease will be eligible, as 153Sm-DOTMP is not expected to cause cardiac dysfunction and is only expected to result in very transient hypocalcemia.
9. A stem cell product collected either by peripheral stem cell mobilization or bone marrow harvest prior to the infusion of CycloSam® must be available, prior to trial entry. A minimum of 2 x 106 CD34+ cells/kg ideal body weight are required.
10. Female subjects of child-bearing potential (defined as premenopausal and capable of becoming pregnant) must have a negative serum pregnancy test at the Screening visit. Females must be surgically sterile, postmenopausal for at least one year prior to Screening (no other medical cause involved) with a Follicle Stimulating Hormone (FSH) level of greater than 40 mIU/mL or must be using a highly effective method of birth control and agree to its use for at least 30 days following the last dose of 153Sm-DOTMP. Highly effective methods of contraceptive are defined as tubal ligation or an approved hormonal contraceptive such as oral contraceptives, patches, implants, injections, rings, or hormonally-impregnated intrauterine device.
11. Male subjects with partners of child-bearing potential must agree to use highly effective methods of contraception for at least 90 days after the last dose of 153Sm-DOTMP.
12. The subject and/or the subject's legally authorized guardian, if the subject is a minor, must acknowledge in writing that informed consent to become a study subject has been obtained, in accordance with institutional policies approved by the U.S. Department of Health and Human Services.
13. Subjects must have previously received effective treatment for their underlying disease and have no potentially curative options available.
14. The concurrent use of hormonal therapies or bisphosphonates is acceptable, provided the latter do not render target lesions invisible on 99mTc bone scan. Subjects will have the option to re-screen up to once more after seven days if they do not initially meet all of the inclusion criteria

Exclusion Criteria:

1. Subject is pregnant or breastfeeding.
2. Subject is sexually active and does not agree to use accepted, effective forms of contraceptive.
3. Subject has received prior radiotherapy to all known areas of current active disease.
4. Subject has a body mass index (BMI) > 50 kg/m2.

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2022-04-05 (Actual); Primary Completion 2024-04-05 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity Rate (DLT) | 42 Days
  The primary endpoint is defined as the DLT rate observed during a 42-day window following administration of 153-Sm-DOTMP for each dose level. DLTs will be defined as any grade 3 or greater hematologic or nonhematologic toxicity, as defined by the National Cancer Institute (NCI) - Common Terminology Criteria for Adverse Events (CTCAE), experienced during a 42 day observation window. The MTD (Maximum Tolerated Dose) will be defined as the dose level that produces a dose limiting toxicity (DLT) rate no greater than 25%.

SECONDARY OUTCOMES:
Bone Tumor Efficacy - Clinical Response Rate | Day 42, 68, 4 months, 8 months, 12 months, 24 months, and 36 months
  Clinical response rate - defined as either SD or a decrease in the size of the tumor by radiographic imaging (which may include CT or MRI) using RECIST v1.1 criteria with the tumor measured in mm by days and months.
Overall Survival | Day 38, 42, 68, 4 months, 6 months, 8 months, 12 months, 24 months, and 36 months
  Overall survival - defined as the time from start of treatment to death due to any cause as measured in days and months
Time to Progression | Day 42, 68, 4 months, 8 months, 12 months, 24 months, and 36 months
  Time to progression - defined as the time from start of treatment to appearance of new lesions or expansion of current lesions by 20% as per RECIST v1.1 criteria in mm of tumor and by days and months
Pain Palliation | Day 38, 42, 68, 4 months, 6 months, 8 months, 12 months, 24 months, and 36 months
  Pain palliation as assessed per the pain VAS as measured in mm of length of a 100 mm Visual Analog Pain Scale by days and months
Safety Based on Number of Treatment Emergent Adverse Events | Day 38, 42, 68, 4 months, 6 months, 8 months, 12 months, 24 months, and 36 months
  Safety based on the number of Treatment Emergent Adverse event (TEAEs), as measured by the number of these events by days and months.

CONTACTS AND LOCATIONS:
Overall Officials: Barry Sugarman, Study Director — QSAM Therapeutics, Inc.
Locations (4):
- United States (4):
  - Clinical Trial Site, Chicago, Illinois
  - Clinical Trial Site, Columbia, Missouri
  - Clinical Trial Site, New Brunswick, New Jersey
  - Clinical Trial Site, Houston, Texas